CLINICAL TRIAL: NCT06419400
Title: A Randomised Controlled Trial to Evaluate the Impact of Supportive Text Messages From GP Practices on Self-reported Symptoms and Inhaler Adherence in Patients With Asthma and/or Chronic Obstructive Pulmonary Disease (COPD) Who Have Been Prescribed a Preventer (Daily) Inhaler (Inhaler Trial)
Brief Title: A Research Study to Explore the Impact of GP Support Via Text Messages to Patients With Asthma and/or COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Accurx (Industry)
Collaborators: Lindus Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Accurx-001
Record Dates: First submitted 2024-05-14; First posted 2024-05-17 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Asthma; COPD
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supportive Text Messagses (Experimental): The intervention group will receive a series of supportive text messages over the 6 month trial period, varying in content and frequency. They will also be asked to provide self reported data on their symptoms and their adherence at 3 points in time (start, mid-point, and end of trial).
  Interventions: Behavioral: Supportive text messages
- Control Group (No Intervention): The control group will receive no supportive text messages over the period of the trial. They will be asked to only provide self reported data on their symptoms and their adherence at 3 points in time (start, mid-point, and end of trial).

INTERVENTIONS:
Behavioral: Supportive text messages — The intervention group will receive a series of supportive text messages over the 6 month trial period, varying in content and frequency.
  Arms: Supportive Text Messagses

SUMMARY:
A 6-month randomised controlled trial to evaluate the impact of text message support on symptom control and inhaler adherence for patients with asthma and/or COPD

DETAILED DESCRIPTION:
This trial will be a 6-month prospective, randomised controlled trial in which the study population is randomly allocated (1:1) to an intervention or control group. The trial is multicentre and is non-blind. All patients in both groups will continue to receive their usual care for the duration of the study. Randomisation will be at the individual level. Participants will be randomly allocated as per a computer-generated randomisation list using a random number generator as part of the Microsoft .NET framework.

This is a behavioural intervention. The intervention will consist of a series of supportive text messages to patients from their GP practice over a 6 month period. The messages will vary in frequency from 2 or 3 in the first weeks of the trial to only 1 or 2 a month in the final months of the trial. The content of the messages will vary; some will contain information about how to use a preventer inhaler, some will emphasise the importance of using it, and some will provide simple reminders to patients to take their inhaler.

All participants will continue to receive their usual care throughout the duration of the study; the text message intervention with be in addition to their usual care.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide informed consent and to comply with the study instructions
2. Male and females age 18 or older
3. Confirmed diagnosis of asthma and/or COPD as recorded in the patient's GP medical record
4. Currently prescribed a preventer inhaler
5. Access to a mobile phone
6. Ability to check text messages on phone
7. Ability to read

Exclusion Criteria:

1. Inability to understand the study procedures
2. Inability or reluctance to provide responses to the study questionnaires
3. Inability to receive and respond to text messages

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6053 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Improved self-reported medication taking as measured by the The Medication Adherence Report Scale (MARS-5) Questionnaire | Baseline to 13 and 26 weeks
  Changes in the MARS-5 Questionnaire

SECONDARY OUTCOMES:
Improved control of asthma symptoms as measured by the Asthma Control Test | Baseline to 13 and 26 weeks (for asthma patients)
  Changes in the Asthma Control Test
A reduction in the interval between patients requesting preventer inhaler prescriptions | Baseline to 13 and 26 weeks
  Reduction in days between consecutive preventer inhaler prescription requests
Difference in emergency admissions | Over 26 weeks
  Differences in the number of emergency admissions between the intervention and control group
Differences in NHS utilisation | Over 26 weeks
  Differences in the utilisation of NHS resources between the intervention and control group

CONTACTS AND LOCATIONS:
Overall Officials: Luke Twelves, Principal Investigator — Lindus Health
Locations (7):
- United Kingdom (7):
  - University Medical Centre, Canterbury, Kent
  - Gravesend Medical Centre, Gravesend, Kent
  - Jubilee Medical Centre, Longfield, Kent
  - Marlowe Park Medical Centre, Rochester, Kent
  - High Oak Surgery, Dudley, West Midlands
  - Lion Health, Stourbridge, West Midlands
  - Wordsley Green Health Centre, Worsley, West Midlands

IPD SHARING:
Plan to Share IPD: No